CLINICAL TRIAL: NCT03991481
Title: A Phase III Multicentre Blinded Randomised Controlled Clinical Non-inferiority Trial of Cryopreserved Platelets vs. Conventional Liquid-stored Platelets for the Management of Surgical Bleeding
Brief Title: The Cryopreserved vs. Liquid Platelets Trial
Acronym: CLIP II
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Australian Red Cross (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZIC-RC/MR002
Record Dates: First submitted 2019-05-09; First posted 2019-06-19 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Surgical Blood Loss; Hemorrhage
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to either: cryopreserved or standard liquid-stored platelets
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Platelets will be allocated to participant by unblinded blood bank staff. The platelets will be supplied by the blood bank with an opaque cover that obscures their method of storage (cryopreserved or liquid-stored), but that retain the original Blood Service information for checking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryopreserved platelets (Experimental): Platelets that have undergone a process to freeze, store and reconstitute platelets, extending their expiry to 2 years
  Interventions: Biological: Cryopreserved platelets
- Liquid-stored platelets (Active Comparator): Platelets that have been liquid stored, with an expiry of 5 days.
  Interventions: Biological: Liquid-stored platelets

INTERVENTIONS:
Biological: Cryopreserved platelets — Platelets that have undergone a process to freeze, store and reconstitute platelets, extending their expiry to 2 years
  Arms: Cryopreserved platelets
Biological: Liquid-stored platelets — Liquid-stored platelets as per standard practice
  Arms: Liquid-stored platelets

SUMMARY:
This trial is a phase III multicentre blinded randomised controlled clinical non-inferiority trial of cryopreserved platelets vs. conventional liquid-stored platelets for the management of surgical bleeding. The aim of the study is to assess the efficacy, safety and cost effectiveness of cryopreserved platelets, compared to conventional liquid-stored platelets, for the management of surgical bleeding. This trial will recruit cardiac surgical patients deemed to be at high risk of surgical bleeding and who may potentially require transfusion of platelets. It is estimated to require 808 high-risk cardiac surgical patients to be recruited, to obtain 202 patients who receive transfused study platelets for surgical bleeding.

DETAILED DESCRIPTION:
For logistic reasons and in order to use this scarce resource optimally, liquid-stored platelets are not stored in smaller hospitals, or in deployed military hospitals. Patients in these hospitals therefore currently have limited or no access to platelet transfusion. Cryopreservation of platelets is a promising technology that would allow smaller hospitals to provide platelet transfusions, reduce overall platelet wastage, and possibly produce better patient outcomes through more effective haemostasis.

This is a phase III multicentre blinded randomised controlled clinical non-inferiority trial of cryopreserved platelets vs. conventional liquid-stored platelets for the management of surgical bleeding. The aim of the study is to assess the efficacy, safety and cost effectiveness of cryopreserved platelets, compared to conventional liquid-stored platelets, for the management of surgical bleeding. This trial will recruit cardiac surgical patients deemed to be at high risk of surgical bleeding and who may potentially require transfusion of platelets. It is estimated to require 808 high-risk cardiac surgical patients to be recruited, to obtain 202 patients who receive transfused study platelets for surgical bleeding. The study will recruit patients in Australian tertiary hospitals.The study hypothesis is that cryopreserved platelets will be at least as effective as conventional liquid-stored platelets in the treatment of active bleeding due to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac surgery patients identified preoperatively as having a high risk of platelet transfusion by either:

   * the ACSePT (Australian Cardiac Surgery Platelet Transfusion (score)) risk prediction tool score ≥1 OR
   * the judgement of the clinicians caring for the patient
2. Written informed consent obtained prior to surgery

Exclusion Criteria:

1. Aged less than 18 years
2. Females of child-bearing age (18- 55 years) who are RhD (Rhesus type D)-negative or whose RhD (Rhesus type D) status is unknown
3. Receipt of platelet transfusion during this hospital admission
4. Deep Vein Thrombosis or Pulmonary Emboli first diagnosed within the preceding 6 months
5. More than one lifetime episode of Deep Vein Thrombosis or Pulmonary Emboli
6. Known inherited or acquired bleeding disorder (e.g. haemophilia, von Willebrand Disease, idiopathic thrombocytopenic purpura, aplastic anaemia, haematological malignancy, chronic liver disease), or any undiagnosed bleeding condition, if (and only if) such a disorder or condition is associated with a significant laboratory abnormality at the time of preoperative screening. i.e.

   * preoperative platelet count <50 000 or
   * INR (International Normalised Ratio) >2 or
   * aPTT (Activated Partial Thromboplastin Time) > 2 x upper limit of normal.
7. Treatment with warfarin, IV heparin or low-molecular weight heparin at "full" therapeutic anticoagulant doses, or other anticoagulant or anti-platelet medications such as factor Xa inhibitors (rivaroxaban, apixaban); factor II inhibitors (dabigatran); adenosine diphosphate receptor inhibitors (clopidogrel, prasugrel, ticagrelor, ticlopidine); glycoprotein IIB/IIIA inhibitors (abciximab, eptifibatide, tirofiban); phosphodiesterase inhibitors (cilostazol); or adenosine reuptake inhibitors (dipyridamole) UNLESS this medication has been discontinued in advance of surgery and its effect allowed to dissipate.
8. Known allergy to dimethylsulphoxide (DMSO)
9. Planned presence of an arterial line and central venous catheter for less than 12 hours postoperatively.
10. Known objection to receipt of human blood components
11. The treating physician believes it is not in the best interest of the patient to be randomised in this trial
12. Previous enrolment during this admission in a clinical trial of a medication or technique thought to influence bleeding, with the exception of any trial of aspirin (i.e. trials involving aspirin are permitted), OR previous enrolment in a clinical trial with a protocol that affects the transfusion of blood products.
13. Previous enrolment in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Volume of post-surgical bleeding in the first 24 hours | First 24 hours from the time of ICU admission
  Volume of post-surgical bleeding in the chest drains after cardiac surgery

SECONDARY OUTCOMES:
Total volume of post-surgical chest drain bleeding | From ICU admission up to removal of drains, death or day 28, whichever occurs first
  Total volume of post-surgical chest drain bleeding, beginning from the time of ICU admission until drain removal
Composite bleeding outcome using the BARC4 criteria | Up to ICU discharge, death or Day 90, whichever occurs first
  Composite bleeding outcome using the Bleeding Academic Research Consortium (BARC4) criteria (intracranial bleeding within 48 hours; reoperation after closure of sternotomy; transfusion of ≥5 Units whole blood or RBCs (red blood cells) within the 48 hour intra- or post-operative period (excluding cell saver blood); chest tube output ≥2 Litres within a 24 hour period)
Number of units of Packed red blood cells transfused | in the first 24 hours after admission to ICU
  Number of units of Packed red blood cells transfused in the first 24 hours after admission to ICU
Total number of units of Packed red blood cells transfused | From operation commencement up to ICU discharge, death or day 90, whichever occurs first
  Total number of units of Packed red blood cells transfused by the time of ICU discharge, including intraoperative transfusion
Occurrence of any one of the following pre-specified potential complications | Up to ICU discharge, death or day 90, whichever occurs first
  Occurrence of any one of the following specified potential complications:
  venous thromboembolism arterial occlusion acute coronary syndrome acute respiratory distress syndrome

OTHER OUTCOMES:
Volume of post-surgical chest drain bleeding | in the first 6, 12, 18, 48 hours, beginning from the time of ICU admission
  Volume of post-surgical chest drain bleeding in the first 6, 12, 18, 48 hours, beginning from the time of ICU admission
Individual elements of the Bleeding Academic Research Consortium (BARC4) composite bleeding outcome | Up to ICU discharge, death or day 90, whichever occurs first
  Individual elements of the Bleeding Academic Research Consortium (BARC4) composite bleeding outcome (intracranial bleeding within 48 hours; reoperation after closure of sternotomy; transfusion of ≥5 Units whole blood or RBC (red blood cells) within the 48 hour intra- or post-operative period (excluding cell saver blood); chest tube output ≥2 Litres within a 24 hour period)
Number of units of blood products | in the first 6, 12, 18, 24, 48 hours*, and at ICU discharge or day 90, death or day 90, whichever occurs first
  Number of units of blood products (Packed red blood cells, plasma, cryoprecipitate, open-label platelets, fibrinogen concentrate, recombinant factor VIIa, prothrombin complex concentrate, whole blood) transfused intraoperatively, in the first 6, 12, 18, 24, 48 hours, and at ICU discharge
Delay between platelet order and commencement of first study platelet infusion | Delay between platelet order and commencement of first study platelet infusion, assessed up to 24 hours
  Delay between platelet order and commencement of first study platelet infusion
Volume of blood in chest drains at the time of ICU admission | From operation commencement up to ICU admission, death or 24 hours, whichever occurs first
  Volume of blood in chest drains at the time of ICU admission
Time to commencement of postoperative aspirin and prophylactic heparin | From ICU admission up to commencement of aspirin and prophylactic heparin, death or day 90, whichever occurs first
  Time to commencement of postoperative aspirin and prophylactic heparin
Volume of fluid resuscitation recorded on the anaesthetic chart | intraoperatively, following ICU admission in the first 6, 12, 18, 24, 48 hours, and at ICU discharge, death or day 90, whichever occurs first
  Volume of fluid resuscitation recorded on the anaesthetic chart intraoperatively, following ICU admission in the first 6, 12, 18, 24, 48 hours, and at ICU discharge
Haemoglobin concentration | results measured on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
  Haemoglobin concentration, on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
Platelet count | results measured on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
  Platelet count on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
Fibrinogen concentration | results measured on day 1 postop and on the last measurement prior to ICU discharge death or day 28, whichever occurs first
  Fibrinogen concentration, on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
INR (International Normalised Ratio) | results measured on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
  INR (International Normalised Ratio) on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
APTT (Activated Partial Thromboplastin Time) | results measured on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
  APTT (Activated Partial Thromboplastin Time) on day 1 postop and on the last measurement prior to ICU discharge, death or day 28, whichever occurs first
Incidence of potential complications of DMSO (preservative used in cryopreserved platelets) | Up to hospital discharge, death or day 90, whichever occurs first
  Incidence of potential complications of DMSO (preservative used in cryopreserved platelets) such as nausea, headache,tachyacrdia, bradycardia, hypertension
Duration of mechanical ventilation | in the first 90 postoperative days for the index admission
  Duration of mechanical ventilation in the first 90 postoperative days for the index admission
Length of postoperative stay in ICU and in hospital | up to ICU and hospital discharge, death or day 90, whichever occurs first
  Length of postoperative stay in ICU and in hospital
Total estimated healthcare cost, incorporating the cost of provision of cryopreserved or liquid-stored platelets | Up to hospital discharge, death or day 90, whichever occurs first
  Total estimated healthcare cost, incorporating the cost of provision of cryopreserved or liquid-stored platelets
mortality at ICU, hospital and 90 days post-enrolment | up to 90 day
  mortality at ICU, hospital and 90 days post-enrolment
ROTEM:EXTEM Clotting time (seconds) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  ROTEM: EXTEM Clotting time (seconds)
ROTEM: EXTEM Clot formation time (seconds) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  ROTEM: EXTEM Clot formation time (seconds)
ROTEM: EXTEM alpha angle (degrees) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  ROTEM:EXTEM alpha angle (degrees)
ROTEM:EXTEM A10 (mm) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  ROTEM:EXTEM A10 (mm)
ROTEM: EXTEM Maximum Clot Firmness (mm) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  ROTEM: EXTEM Maximum Clot Firmness (mm)
ROTEM: EXTEM Lysis Index 30 min after CT (LI30) (%) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  ROTEM: EXTEM Lysis Index 30 min after CT (LI30) (%)
TEG: Standard (Kaolin) Reaction (R) time (seconds) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  TEG: Standard (Kaolin) Reaction (R) time (seconds)
TEG: Standard (Kaolin) Clot formation (K) time (seconds) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  TEG: Standard (Kaolin) Clot formation (K) time (seconds)
TEG: Standard (Kaolin) Alpha angle (degrees) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  TEG: Standard (Kaolin) Alpha angle (degrees)
TEG: Standard (Kaolin) Maximum amplitude (mm) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  TEG: Standard (Kaolin) Maximum amplitude (mm)
TEG: Standard (Kaolin) Lysis at 30 mins (LY30) (%) | Results before and after last study platelet transfusion (where performed) through study completion up to day 28.
  TEG: Standard (Kaolin) Lysis at 30 mins (LY30) (%)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reade, Study Chair — ANZIC-Research Centre; Australian Defence Force, University of Queensland,
Locations (6):
- Australia (6):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Yes
At the completion of the study, at the discretion of the trial Management Committee and Monash University, an extract of the trial data without any patient identifiers may be made available on a case-by-case basis to investigators from reputable research organisations with a defined protocol and analysis plan, using the principles to protect patient anonymity described by the UK Medical Research Council. In accordance with the Australian & New Zealand Intensive Care Society Clinical Trials Group (ANZICS CTG) Terms of Reference for an endorsed trial, the CTG Chair must approve sharing of data with any third party, manuscripts derived from shared data must be submitted for CTG endorsement prior to publication and must acknowledge the role of the CTG in the original study, and a copy of the published manuscript must be provided to the CTG office.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data availability will begin 9 months after publication of the individual patient data meta-analysis combining both trial results, and end 36 months after this publication.
Access Criteria: Submissions to use data with investigators from reputable research organisations with a defined protocol and analysis plan, using the principles to protect patient anonymity described by the UK Medical Research Council.

REFERENCES:
- [Derived] Reade MC, Marks DC, Howe BD, Bailey MJ, Bannon PG, Eastwood GM, French CJ, Gattas DJ, Higgins AM, Holley AD, Hu RT, Irving DO, Johnson L, McGuinness SP, McQuilten ZK, Royse AG, Smith JA, Weinberg L, Wood EM; Cryopreserved vs Liquid Platelets II (CLIP-II) Investigators, the Australian and New Zealand Intensive Care Society Clinical Trials Group, the Australian and New Zealand College of Anaesthetists Clinical Trials Network, and the Australasian Society of Car; Cryopreserved vs Liquid Platelets II (CLIP-II) Investigators, the Australian and New Zealand Intensive Care Society Clinical Trials Group, the Australian and New Zealand College of Anaesthetists Clinical Trials Network, and the Australasian Society of Cardiac and Thoracic Surgeons. Cryopreserved vs Liquid-Stored Platelets for the Treatment of Surgical Bleeding: The CLIP-II Randomized Noninferiority Clinical Trial. JAMA. 2025 Dec 8:e2523355. doi: 10.1001/jama.2025.23355. Online ahead of print. PMID 41360717
- [Derived] Reade MC, Marks DC, Howe B, McGuinness S, Parke R, Navarra L, Charlewood R, Johnson L, McQuilten Z; CLIP-II and CLIPNZ-II Investigators.; CLIP-II and CLIPNZ-II Investigators. Cryopreserved platelets compared with liquid-stored platelets for the treatment of surgical bleeding: protocol for two multicentre randomised controlled blinded non-inferiority trials (the CLIP-II and CLIPNZ-II trials). BMJ Open. 2022 Dec 20;12(12):e068933. doi: 10.1136/bmjopen-2022-068933. PMID 36600425